CLINICAL TRIAL: NCT04868617
Title: ATTRACT-I: A Randomized Controlled Clinical Investigation Evaluating a Flat Ostomy Barrier With A Novel Skin Protection Technology
Brief Title: A Randomized Controlled Clinical Investigation Evaluating a Flat Ostomy Barrier With A Novel Skin Protection Technology
Acronym: CP338
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP338
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Peristomal Skin Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): The non-CE marked test product is a stoma product based on the flat SenSura® Mio 1-piece (1-pc) and the flat 2-piece with mechanical coupling (2-pc MC) product that includes a novel skin protective layer in the baseplate.
  Interventions: Device: ATTRACT-I
- SenSura® Mio Comparator - Standard of Care (Active Comparator): The following comparator products will be used in this investigation:
  * SenSura® Mio 1-piece (1-pc) flat, Midi bag with normal outlet and
  * SenSura® Mio 2-piece with mechanical coupling (2-pc MC) flat, Maxi or Midi bag with normal outlet
  Interventions: Device: ATTRACT-I

INTERVENTIONS:
Device: ATTRACT-I — The aim of this investigation is to evaluate the performance and safety of an ostomy baseplate with a novel skin protection technology and its ability to reduce peristomal skin complications compared to SenSura® Mio. The subject will be randomized to either test product or comparator at enrollment. The subject will wear the test product for approximately 35 days and then cross-over to the comparator (or vice-versa) for approximately 35 days. At each baseplate change, the subject will answer questions about their skin, and take pictures of their stoma and used baseplate. They will also answer quality of life questionnaires at each study visit.

SUMMARY:
This investigation is a randomized, controlled, open-label, comparative, cross-over, multicenter investigation, with two test periods. In total, 82 subjects will be included and randomized, and each subject will have three test visits overseen by the Principal Investigator, or designee. Each subject will be enrolled for 2 × 35 -1/+3 days in total for the entire investigation, thus approximately 70 days. The subjects will test the non-CE marked test product and the comparator product in randomized order.

DETAILED DESCRIPTION:
People with intestinal stomas have, despite development of better stoma products, problems with leakage induced peristomal skin complications which influence quality of life negatively. In fact, the primary cause of peristomal skin complication development is due to leakage of ostomy effluents under the adhesive barrier. Some of the common clinical signs of peristomal skin complications include pain, itching, burning, discoloration, bleeding, and wounds . To overcome this, Coloplast A/S has developed a new baseplate which is comprised of a protective layer.

This investigation is a randomised, controlled, open-label, comparative, cross-over, multicentre investigation, with two test periods. In total 82 subjects will be included and randomised, and each subject will have at least three test visits overseen by the Principal Investigator, or designee. Each subject will be enrolled for 2 × 35 -1/+3 days; thus approximately 70 days. The subjects will test the non-CE marked investigational product and the comparator product in a randomised order.

Before the test periods, the subjects are invited for a screening visit (V0). Subjects will be consented prior to any study procedures. Once consented, during their participation, the subjects will complete three study visits (V1, V2 and V3). The visits can be at the Principal Investigators clinic or in the subject's home. In rare cases (i.e. global pandemic), visits can be done remotely via video conference. In addition, the Principal Investigator, or designee, will call the subjects four times during the course of the investigation to inquire if the subject has had any issues or concerns.

During the test visits the subject will complete a quality of life questionnaire and discuss/record any adverse events or device deficiencies. The subject will also be asked about the use and handling of the product, and their preference.

At every baseplate change the subjects will be asked to take photos of their stoma/peristomal skin and the backside (adhesive side) of the used product. The photos will be taken with a smartphone using the Coloplast Clinical Trial App. The subject will also be asked to complete a questionnaire about their peristomal skin condition.

Coloplast will provide both the investigational product and the comparator product for all subjects.

If a subject experiences a problem with the investigational product during the investigation, he/she should contact the investigator for advice. Subjects that cannot complete a test period with the test product may choose to use their own product (i.e., SenSura® Mio) for the remainder of the test period. However, this must be documented by the Principal Investigator.

The duration of the test periods (35 -1/+3 days) and number of visits should be adequate to assess data on the skin condition of the subjects. The investigational products are tested for 35 -1/+3 days in each study period to ensure that the skin will have time to adjust to new conditions, reach a steady state, and for the subjects to test the product for an adequate number of days to give a thorough evaluation of the products.

To account for a possible carry-over effect, the steady state period of the treatment period begins after two weeks of product use. It is anticipated that the skin will have adapted to the new product after two weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written consent to participate by signing the Informed Consent Signature Form
2. Is at least 18 years of age and have full legal capacity
3. Has an ileostomy or colostomy with consistent liquid fecal output (6-7 Bristol scale.
4. Is currently using a SenSura® Mio flat product with open bag.
5. Has had the ostomy for at least 90 days.
6. Can use an ostomy product with a max cut size of 45 mm (1-piece) or 38 mm (2-piece).
7. Has experienced leakage** under the baseplate at least three times within the last fourteen days.

   **Leakage defined as output/seeping under the baseplate (see appendix 7)
8. Has experienced symptoms of peristomal skin complications such as itching, burning, or pain in the peristomal area within the last fourteen days. **

   ** Proper training of the PI and nurses in how to ask the subject about these symptoms is essential.
9. Is able to handle the electronic diary (questionnaire/photo) themselves. If needed, a trained spouse or caretaker is allowed to assist.
10. Is able to handle (apply, remove, cut, etc.) the product themselves.
11. Understands that any barrier products (film, cream, spray, wipes etc.) are not permissible during the investigation, and is willing to not use these accessories during the investigation.
12. Is willing and suitable (determined by the Principal Investigator or designee) to use a flat custom cut one-piece open or two-piece open product during the investigation.
13. Is willing to change the product (1-piece) or baseplate (2-piece) at least every fourth days.

Exclusion Criteria:

1. Is currently receiving or have within the past 60 days received radio-and/or chemotherapy.

   - low doses radio- and/or chemotherapy (assessed by Principal Investigator) is allowed for other indications than cancer.
2. Is currently receiving or have within the past 30 days received topical steroid treatment in the peristomal skin area, e.g., lotion or spray.

   * Low dose systemic steroid treatment (e.g., inhalation) assessed by the investigator are allowed.
   * Other systemic steroid treatment (e.g., injection or tablet) are not allowed.
3. Is breastfeeding.
4. Is pregnant based on urine pregnancy test.
5. Has known hypersensitivity towards any of the products used in the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Karlsmark, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product - the Non-CE Marked Product, Then Standard of Care: Participants first received the test product (the non-Conformité Européene marked product) for 35 -1/+3 days. Then there was a cross-over and the participants received the standard of care (the Conformité Européene marked product) for 35 -1/+3 days. There was no 'Washout period'
  The test product used was the non-Conformité Européene marked product which was a stoma product based on the flat SenSura® Mio 1-piece and the flat 2-piece with mechanical coupling product that includes a novel skin protective layer in the baseplate.
  The following standard of care products (the Conformité Européene marked product) was used in this investigation:
  * SenSura® Mio 1-piece flat, Midi bag with normal outlet and
  * SenSura® Mio 2-piece with mechanical coupling flat, Maxi or Midi bag with normal outlet
- Standard of Care, Then the Test Product - the Non-CE Marked Product: Participants first received standard of care (the Conformité Européene marked product) for 35 -1/+3 days. Then there was a cross-over and the participants received the test product (the non-Conformité Européene marked comparator product) for 35 -1/+3 days. There was no 'Washout period'.
  The test product used was the non-Conformité Européene marked product which was a stoma product based on the flat SenSura® Mio 1-piece and the flat 2-piece with mechanical coupling product that includes a novel skin protective layer in the baseplate.
  The following standard of care products (the Conformité Européene marked product) was used in this investigation:
  * SenSura® Mio 1-piece flat, Midi bag with normal outlet and
  * SenSura® Mio 2-piece with mechanical coupling flat, Maxi or Midi bag with normal outlet
Period: Overall Study
Arm/Group | Test Product - the Non-CE Marked Product, Then Standard of Care | Standard of Care, Then the Test Product - the Non-CE Marked Product
Started | 42 | 41
Completed | 38 | 41
Not Completed | 4 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Device deficiency | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population Baseline Measures: The non-CE marked test product is a stoma product based on the flat SenSura® Mio 1-piece (1-pc) and the flat 2-piece with mechanical coupling (2-pc MC) product that includes a novel skin protective layer in the baseplate.
  Arm 1: Participants first received the non-Conformité Européene marked test product for 35 -1/+3 days. Then there was a cross-over and the participants received the Conformité Européene comparator product (standard of care) for 35 -1/+3 days.
  Arm 2: Participants first received the Conformité Européene marked comparator product for 35 -1/+3 days. Then there was a cross-over and the participants received the non-Conformité Européene test product for 35 -1/+3 days.
Arm/Group | Total ITT Population Baseline Measures
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 5
  Sweden | 11
  Norway | 13
  Germany | 22
  United Kingdom | 28
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (6.5)
Height (cm) [Mean (Standard Deviation); unit: cm] | 172.2 (10.1)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 83.8 (20.1)
Stoma age (Years since surgery) [Mean (Standard Deviation); unit: years] | 11.2 (10.4)
Type of stoma; ileostomy / colostomy [Count of Participants; unit: Participants]
  Ileostomy | 53
  Colostomy | 26
Stoma diameter (mm) [Mean (Standard Deviation); unit: mm] | 29.2 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: The Peristomal Skin Condition Measured by the Decision Tree Score (Scale From 0-3)
Description: The peristomal skin condition measured by the Decision Tree Score on baseplate level at steady state (scale from 0-3). Higher score means worse outcome
Time Frame: after 5 weeks
Population: Intention to treat (ITT)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Test Product: The non-Conformité Européene marked test product is a stoma product based on the flat SenSura® Mio 1-piece and the flat 2-piece with mechanical coupling product that includes a novel skin protective layer in the baseplate.
  Arm 1: Participants first received the non-Conformité Européene marked test product for 35 -1/+3 days. Then there was a cross-over and the participants received the Conformité Européene comparator product (standard of care) for 35 -1/+3 days.
  Arm 2: Participants first received the Conformité Européene marked comparator product for 35 -1/+3 days. Then there was a cross-over and the participants received the non-Conformité Européene test product for 35 -1/+3 days.
- Standard of Care: The following comparator products (standard of care) will be used in this investigation:
  * SenSura® Mio 1-piece flat, Midi bag with normal outlet and
  * SenSura® Mio 2-piece with mechanical coupling flat, Maxi or Midi bag with normal outlet
  Arm 1: Participants first received the non-Conformité Européene marked test product for 35 -1/+3 days. Then there was a cross-over and the participants received the Conformité Européene comparator product (standard of care) for 35 -1/+3 days.
  Arm 2: Participants first received the Conformité Européene marked comparator product for 35 -1/+3 days. Then there was a cross-over and the participants received the non-Conformité Européene test product for 35 -1/+3 days.
Arm/Group | Test Product | Standard of Care
Number analyzed (Participants) | 79 | 79
score on a scale | 1.8 [1.6 to 2.0] | 2.0 [1.8 to 2.2]
Statistical Analysis 1: Comparison: Test Product vs Standard of Care; Test type: Superiority; p = 0.015, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to -0.03]

2. Secondary Outcome: Health-related Quality of Life (Scale 0-30)
Description: A health-related quality of life measured by the DLQI score evaluated at the end of each test period (scale from 0-30, the higher the score, the worse the QoL for the participant)
Time Frame: 5 weeks
Population: Intention to treat (ITT)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Standard of Care: The following comparator products will be used in this investigation:
  * SenSura® Mio 1-piece (1-pc) flat, Midi bag with normal outlet and
  * SenSura® Mio 2-piece with mechanical coupling (2-pc MC) flat, Maxi or Midi bag with normal outlet
  ATTRACT-I: The aim of this investigation is to evaluate the performance and safety of an ostomy baseplate with a novel skin protection technology and its ability to reduce peristomal skin complications compared to SenSura® Mio. The subject will be randomized to either test product or comparator at enrollment. The subject will wear the test product for approximately 35 days and then cross-over to the comparator (or vice-versa) for approximately 35 days. At each baseplate change, the subject will answer questions about their skin, and take pictures of their stoma and used baseplate. They will also answer quality of life questionnaires at each study visit.
Arm/Group | Test Product | Standard of Care
Number analyzed (Participants) | 79 | 79
score on a scale | 3.2 [2.4 to 4.1] | 4.0 [3.2 to 4.8]
Statistical Analysis 1: Comparison: Test Product vs Standard of Care; Test type: Superiority; p = 0.035, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.5 to -0.1]

ADVERSE EVENTS:
Time Frame: Each subject was enrolled for 2x for 35 -1/+3 days in total for the entire investigation, thus approximately 70 days.
Description: The relationship to the investigational or comparator product were collected. The safety population constituted the subjects who had given informed consent and were 89 participants. The participants in each arm represent an adverse event reported that was either: "Not Related", "Unlikely Related", "Possibly Related", "Probably Related" or "Causal relationship" to the Non-Conformité Eurppéene Marked Product or the Conformité Européene Marked product.
Groups:
- Standard of Care: The following Conformité Européene marked comparator product (standard of care) will be used in this investigation:
  * SenSura® Mio 1-piece flat, Midi bag with normal outlet and
  * SenSura® Mio 2-piece with mechanical coupling flat, Maxi or Midi bag with normal outlet
  Arm 1: Participants first received the non-Conformité Européene marked test product for 35 -1/+3 days. Then there was a cross-over and the participants received the Conformité Européene comparator product (standard of care) for 35 -1/+3 days.
  Arm 2: Participants first received the Conformité Européene marked comparator product for 35 -1/+3 days. Then there was a cross-over and the participants received the non-Conformité Européene test product for 35 -1/+3 days.
- Total Safety Population: This arm group constitutes the safety population
Arm/Group | Test Product | Standard of Care | Total Safety Population
All-Cause Mortality (participants affected / at risk) | 1/85 | 0/79 | 1/89
Serious Adverse Events (participants affected / at risk) | 1/85 | 1/79 | 2/89
Other Adverse Events (participants affected / at risk) | 21/85 | 19/79 | 29/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (N=85) | Standard of Care (N=79) | Total Safety Population (N=89)
Knee injury meniscusresection (Surgical and medical procedures) | 0 | 1 | 1
Multi organ failure (General disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=85) | Standard of Care (N=79) | Total Safety Population (N=89)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Eye disorders (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (8) | 5 (6) | 7 (14)
General disorders/adm site conditions (General disorders) | 1 (1) | 1 (1) | 2 (2)
Infections and infestations (Infections and infestations) | 3 (3) | 3 (3) | 5 (6)
Injury poisoning /procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal/connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 5 (6)
Nervous system disorders (Nervous system disorders) | 2 (2) | 4 (4) | 6 (6)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory thoracic/mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2) | 6 (8)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 7 (13) | 5 (8) | 12 (21)
Surgical and medical procedure (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the investigation, may be communicated by abstracts, posters, or oral presentations provided that opportunity is given for sponsor to discuss the contents and any conclusions drawn, before the abstract, paper, or visual presentations are finalized. Sponsor will undertake to comment on the draft documents within 30 working days of receipt, but the final decision on the contents and format of the publication from the conclusions drawn, will remain with the authors.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT04868617/Prot_SAP_000.pdf